CLINICAL TRIAL: NCT07197333
Title: Mean Platelet Volume and Platelet Distribution Width as Early Indicators of Deep Vein Thrombosis and Prognostic Markers in Mechanically Ventilated Intensive Care Unit Patients
Brief Title: Early Platelet Indices as Biomarkers of Deep Vein Thrombosis and Prognostic Markers in Mechanically Ventilated ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Roiea Abd El Reheem Aref, resident at the Critical Care Medicine department, Assiut University
Other Study IDs: Predictors of DVT
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Platelet Distribution Width; Mean Platelet Volume
Keywords: platelet distribution width; mean platelet volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult critically ill patients aged ≥18 years admitted to the ICU of Assiut University Hospital who r: The population will consist of mechanically ventilated ICU patients, a group at particularly high risk of thrombotic events due to immobility, systemic inflammation, and sedation, which limit symptom reporting. Eligible participants must be adults (>18 years) who remain intubated for ≥48 hours.

SUMMARY:
This prospective observational study aims to evaluate the role of mean platelet volume (MPV) and platelet distribution width (PDW) as early indicators of deep vein thrombosis (DVT) and as prognostic markers in mechanically ventilated Intensive Care Unit (ICU) patients.

DETAILED DESCRIPTION:
The study will be conducted at the Critical Care Unit of Assiut University Hospital and will recruit 100 mechanically ventilated patients. Deep venous thrombosis (DVT) remains a major challenge in ICU patients due to the difficulty in clinical detection. Conventional tools such as Doppler ultrasound and D-dimer testing have significant limitations, creating a need for cost-efficient, accessible biomarkers. MPV and PDW are promising markers of platelet activation and variability, both of which play central roles in thrombus formation. These indices are routinely included in complete blood count (CBC) tests, making them widely accessible.

The study will explore whether elevated MPV and PDW values at ICU admission and during follow-up are associated with higher incidence of DVT and increased ICU mortality. Patients will undergo baseline investigations, followed by repeated platelet measurements every 48 hours until ICU discharge or death. Doppler ultrasound assessments will be done on Day 5-7 or earlier if symptoms suggest thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years

Admitted to ICU at Assiut University Hospital

Mechanically ventilated for ≥48 hours

Exclusion Criteria:

* Known hematological malignancy or platelet disorders

Recent platelet transfusion within 7 days

Known pre-existing deep vein thrombosis

Previous anticoagulation treatment prior to ICU admission

Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he population will consist of mechanically ventilated ICU patients, a group at particularly high risk of thrombotic events due to immobility, systemic inflammation, and sedation, which limit symptom reporting. Eligible participants must be adults (>18 years) who remain intubated for ≥48 hours. Patients with confounding conditions such as hematological malignancies, congenital platelet disorders, recent platelet transfusions, pre-existing DVT, anticoagulation therapy prior to ICU admission, or pregnancy will be excluded. This selection creates a homogeneous population highly vulnerable to DVT, ideal for assessing the predictive value of MPV and PDW.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DVT during ICU stay | one day
  Percentage of patients developing DVT as confirmed by Doppler ultrasound during ICU admission

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Xu Z, Li Z, et al. Mean platelet volume and platelet distribution width as prognostic markers in critically ill patients with sepsis. J Crit Care. 2019;50:213-219. doi:10.1016/j.jcrc.2018.12.003